CLINICAL TRIAL: NCT03473431
Title: A Pilot Study of a Single Infusion of Ketamine in Relief of Depressive Symptoms of Elderly Patients With Visual Impairment.
Brief Title: Effect of Ketamine in Depressive Symptoms of Elderly Patients With Visual Impairment.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Instituto de Seguridad y Servicios Sociales de los Trabajadores del Estado (Other Government)
Responsible Party: Principal Investigator, Dulce Maria Rascon Martinez, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IMexicanoSS
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Depression in Old Age; Ketamine
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, dose-controlled follow-up study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ketamine (Experimental): single infusion of 0.5 mg / kg ketamine
  Interventions: Drug: Ketamine
- control (Sham Comparator): physiological solution at 0.9 % with the same physical characteristics of ketamine solution,
  Interventions: Other: control

INTERVENTIONS:
Drug: Ketamine — single infusion of 0.5 mg / kg ketamine
  Arms: ketamine
Other: control — physiological solution at 0.9 % with the same physical characteristics of ketamine solution,
  Arms: control

SUMMARY:
the prevalence of depression in elderly is from 4 to 30% and is associated with a lower quality of life mayor medical comorbidity, and increased mortality. Although there are various treatments for depression in the elderly, the study of interventions in resistant depression is limited and there are few reports of the efficacy and safety profile of alternative interventions such as ketamine in the elderly. The final objective of the present study is to report the effects of a single infusion of ketamine on the depressive symptoms in patients undergoing ophthalmologic surgery

DETAILED DESCRIPTION:
The final objective of the present study is to report the effects of a single infusion of 0.5 mg / kg ketamine in infusion on depressive symptoms assessed using the scale Yesavage's abbreviated Geriatric Depression Scale.

This is a randomized double-blind follow-up study in patients over 60 years of age with ocular pathology who required ophthalmological surgery with retrobulbar block and conscious sedation with ketamine. The sample consisted of two groups: a control group and an experimental group with ketamine. The dose used for the study was 0.5mg / kg in slow infusion for two hours. In both groups the Yesavage's questionnaire was applied at three different times; Basally, at the end of the recovery and at 24 hours after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 60 years or older who due to the severity of visual disability required to be operated on for eye surgery using retrobulbar block
* Intraocular pressure <20 mm Hg and
* ASA functional capacity from I to III

Exclusion Criteria:

* Previous antidepressants medications
* Cognitive impairment was found according to the Short Portable Mental Status Questionnaire (SPMSQ) assessment
* In case of a history of psychosis, schizophrenia, nephropathy
* They had a history of difficulties to control arterial blood pressure, uncontrolled hepatic disorders or had a history of adverse response to ketamine according clinical records

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | two hours and 24 hours after the ketamine infusion
  Change in the total score in a scale for Geriatric Depression the "Geriatric Depression Scale. " It will be consider as an outcome the total score. The scale have a maximun score of 15 and minimum of 0. Higher values are considered a worse outcome.

SECONDARY OUTCOMES:
Depression rate | two hours and 24 hours after the ketamine infusion
  change in the percentage of patients with criteria for depression based on cutting point of 5 scale

CONTACTS AND LOCATIONS:
Overall Officials: DULCE RASCON MARTINEZ, M.D, Principal Investigator — imss
Locations (1):
- Centro Medico Nacional Siglo XXI. UMAE Hospital de Especialidades, Mexico City, Mexico City, Mexico

REFERENCES:
- [Background] Andrade C. Ketamine for Depression, 1: Clinical Summary of Issues Related to Efficacy, Adverse Effects, and Mechanism of Action. J Clin Psychiatry. 2017 Apr;78(4):e415-e419. doi: 10.4088/JCP.17f11567. PMID 28448702
- [Background] Arandjelovic K, Eyre HA, Lavretsky H. Clinicians' Views on Treatment-Resistant Depression: 2016 Survey Reports. Am J Geriatr Psychiatry. 2016 Oct;24(10):913-7. doi: 10.1016/j.jagp.2016.05.010. Epub 2016 May 18. PMID 27591914
- [Background] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Background] Collins PY, Patel V, Joestl SS, March D, Insel TR, Daar AS; Scientific Advisory Board and the Executive Committee of the Grand Challenges on Global Mental Health; Anderson W, Dhansay MA, Phillips A, Shurin S, Walport M, Ewart W, Savill SJ, Bordin IA, Costello EJ, Durkin M, Fairburn C, Glass RI, Hall W, Huang Y, Hyman SE, Jamison K, Kaaya S, Kapur S, Kleinman A, Ogunniyi A, Otero-Ojeda A, Poo MM, Ravindranath V, Sahakian BJ, Saxena S, Singer PA, Stein DJ. Grand challenges in global mental health. Nature. 2011 Jul 6;475(7354):27-30. doi: 10.1038/475027a. No abstract available. PMID 21734685
- [Background] Fond G, Loundou A, Rabu C, Macgregor A, Lancon C, Brittner M, Micoulaud-Franchi JA, Richieri R, Courtet P, Abbar M, Roger M, Leboyer M, Boyer L. Ketamine administration in depressive disorders: a systematic review and meta-analysis. Psychopharmacology (Berl). 2014 Sep;231(18):3663-76. doi: 10.1007/s00213-014-3664-5. Epub 2014 Jul 20. PMID 25038867
- [Background] George D, Galvez V, Martin D, Kumar D, Leyden J, Hadzi-Pavlovic D, Harper S, Brodaty H, Glue P, Taylor R, Mitchell PB, Loo CK. Pilot Randomized Controlled Trial of Titrated Subcutaneous Ketamine in Older Patients with Treatment-Resistant Depression. Am J Geriatr Psychiatry. 2017 Nov;25(11):1199-1209. doi: 10.1016/j.jagp.2017.06.007. Epub 2017 Jun 13. PMID 28739263
- [Background] Han Y, Chen J, Zou D, Zheng P, Li Q, Wang H, Li P, Zhou X, Zhang Y, Liu Y, Xie P. Efficacy of ketamine in the rapid treatment of major depressive disorder: a meta-analysis of randomized, double-blind, placebo-controlled studies. Neuropsychiatr Dis Treat. 2016 Nov 3;12:2859-2867. doi: 10.2147/NDT.S117146. eCollection 2016. PMID 27843321
- [Background] Martinez de la Iglesia, J., Onis Vilches Ma, C., Duenas Herrero, R., Albert Colomer, C., Aguado Taberne, C., & Luque Luque, R. (2002). The Spanish version of the Yesavage abbreviated questionnaire (GDS) to screen depressive dysfunctions in patients older than 65 years. [Spanish]. MEDIFAM - Revista de Medicina Familiar Y Comunitaria, 12(10), 620-630
- [Background] Stek ML, Vinkers DJ, Gussekloo J, van der Mast RC, Beekman AT, Westendorp RG. Natural history of depression in the oldest old: population-based prospective study. Br J Psychiatry. 2006 Jan;188:65-9. doi: 10.1192/bjp.188.1.65. PMID 16388072
- [Background] Volkert J, Schulz H, Harter M, Wlodarczyk O, Andreas S. The prevalence of mental disorders in older people in Western countries - a meta-analysis. Ageing Res Rev. 2013 Jan;12(1):339-53. doi: 10.1016/j.arr.2012.09.004. Epub 2012 Sep 19. PMID 23000171